CLINICAL TRIAL: NCT00001589
Title: Comparison of Asymptomatic Carotid Atherosclerosis Between Frequent and Infrequent Blood Donors
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 970113; 97-CC-0113
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2002-05

CONDITIONS: Carotid Atherosclerosis; Myocardial Infarction
Keywords: Ferritin; Atherosclerosis; Myocardial Infarction; Blood Donors; Low Density Lipoprotein; Asymptomatic Carotid Atherosclerosis
MeSH Terms: conditions — Carotid Artery Diseases; Myocardial Infarction; Atherosclerosis

SUMMARY:
Iron has been proposed to contribute to atherogenesis in humans by facilitating the oxidation of lipoproteins. This observational study will evaluate the association between frequency of blood donation - expected to be associated with relatively reduced body iron stores in frequent donors - and carotid atherosclerosis. The primary outcome variable will be whether the presence and extent of asymptomatic carotid atherosclerosis as measured by ultrasound is greater in infrequent (less than or equal to 1 donations/year greater than or equal to 5 years) vs. frequent (greater than or equal to 4 donations/year greater than or equal to 5 years) blood donors. Body iron stores, lipid and hemostatic parameters, nitric oxide formation, inflammatory parameters, and markers of vascular oxidative stress will be analyzed as secondary outcome measures. Laboratory analysis and ultrasound testing will be performed blinded to the patient's phlebotomy and iron status. Sixty frequent (n=40 males greater than 40 y/o, n=20 females greater than 50 y/o) and 60 infrequent (n=40 males greater than 40 y/o, n=20 females greater than 50 y/o) blood donors will be recruited for this study from the Department of Transfusion Medicine, W. G. Magnuson Clinical Center. All donors will be assessed for study eligibility and cardiovascular risks during the screening visit. The presence of atherosclerotic lesions by carotid ultrasound and secondary outcome parameters will be assessed during a second visit.

DETAILED DESCRIPTION:
Iron has been proposed to contribute to atherogenesis in humans by facilitating the oxidation of lipoproteins. This observational study will evaluate the association between frequency of blood donation - expected to be associated with relatively reduced body iron stores in frequent donors - and carotid atherosclerosis. The primary outcome variable will be whether the presence and extent of asymptomatic carotid atherosclerosis as measured by ultrasound is greater in infrequent (less than or equal to 1 donations/year greater than or equal to 5 years) vs. frequent (greater than or equal to 4 donations/year greater than or equal to 5 years) blood donors. Body iron stores, lipid and hemostatic parameters, nitric oxide formation, inflammatory parameters, and markers of vascular oxidative stress will be analyzed as secondary outcome measures. Laboratory analysis and ultrasound testing will be performed blinded to the patient's phlebotomy and iron status. Sixty frequent (n=40 males greater than 40 y/o, n=20 females greater than 50 y/o) and 60 infrequent (n=40 males greater than 40 y/o, n=20 females greater than 50 y/o) blood donors will be recruited for this study from the Department of Transfusion Medicine, W. G. Magnuson Clinical Center. All donors will be assessed for study eligibility and cardiovascular risks during the screening visit. The presence of atherosclerotic lesions by carotid ultrasound and secondary outcome parameters will be assessed during a second visit.

ELIGIBILITY:
INCLUSION CRITERIA:

Age greater than or equal to 40 years for males and greater than or equal to 50 years for females.

Standard eligibility criteria for blood donation, per guidelines established by the Food and Drug Administration and the American Association of Blood Banks.

Ability to provide consent after full information is provided.

EXCLUSION CRITERIA:

Pregnancy or lactation.

Patients with clinically significant dementia or psychiatric disturbances, including alcohol and substance abuse.

Presence of the following American Heart Association cardiovascular risks: diabetes mellitus, hypertension (systolic greater than 140 mmHg, diastolic greater than 90 mmHg), smoking (greater than 10 cigarettes/day), high density lipoprotein cholesterol less than 35 mg/dL, hyperlipidemia (total cholesterol greater than 240 mg/dL), family history of premature coronary heart disease.

Anticoagulant, thrombolytic, hemorrheologic and/or antiplatelet agents (within the last 10 days).

Any other condition or therapy which in the opinion of the investigators may pose a risk to the patient or confound the results of the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 120
Dates: Start 1997-04; Study Completion 2002-05

CONTACTS AND LOCATIONS:
Locations (1):
- Warren G. Magnuson Clinical Center (CC), Bethesda, Maryland, United States

REFERENCES:
- [Background] Fuster V. Lewis A. Conner Memorial Lecture. Mechanisms leading to myocardial infarction: insights from studies of vascular biology. Circulation. 1994 Oct;90(4):2126-46. doi: 10.1161/01.cir.90.4.2126. PMID 7718033
- [Background] Rader DJ, Hoeg JM, Brewer HB Jr. Quantitation of plasma apolipoproteins in the primary and secondary prevention of coronary artery disease. Ann Intern Med. 1994 Jun 15;120(12):1012-25. doi: 10.7326/0003-4819-120-12-199406150-00008. PMID 8185133
- [Background] Kannel WB. Clinical misconceptions dispelled by epidemiological research. Circulation. 1995 Dec 1;92(11):3350-60. doi: 10.1161/01.cir.92.11.3350. PMID 7586324